CLINICAL TRIAL: NCT05425121
Title: Effects of Core Stability Exercises With Surface Electromyography Biofeedback on Postural Stability and Sensory Integration of Balance in Patients With Mechanical Low Back Pain
Brief Title: Core Stability Exercises With Surface Electromyography Biofeedback in Patients With Mechanical Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCRS&AHS/22/1105
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Low Back Pain
Keywords: Low back pain; Postural stability; Sensory integration of balance; Surface Electromyography Biofeedback
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to control Group A (Core stability training protocol ) or Interventional Group B(core stability training protocol with surface electromyography biofeedback protocol) for the whole duration of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stability protocol (Active Comparator): Participants in this group will undergo core stability exercise program . Each exercise plan will be progressively increased.
  Interventions: Procedure: Core stability exercises
- Core Stability with surface electromyography biofeedback (Experimental): Participants in this group will undergo core stability exercise program with surface electromyography biofeedback. Each exercise plan will be progressively increased with application of surface electromyography biofeedback.
  Interventions: Procedure: Core stability exercises; Device: Biofeedback training

INTERVENTIONS:
Procedure: Core stability exercises — The intervention in the control group will core stability exercises for different back muscles and strengthening exercises of Gluteal Muscles.
Device: Biofeedback training — EMG biofeedback training will be administered to the participants in combination with core stability exercise training.
  Arms: Core Stability with surface electromyography biofeedback

SUMMARY:
This study will be conducted on patients of mechanical low back pain. Surface electromyography biofeedback driven core stability protocol will be given to experimental group and the control group will be treated with core stabilization regimen. Then it will compare the effects of surface electromyography biofeedback with core stability on postural stability and sensory integration of balance .

DETAILED DESCRIPTION:
Low back pain is very common musculoskeletal condition involving lumbar spine .it is almost affecting 80 % of world's population. Mostly it is self-limiting but it is episodic in nature.it is not an isolated problem it is usually associated with social occupational stresses and psychological issues.it is significantly associated with severe disruption in functional disability morbidity. Postural control involves information processing from sensory stimuli derived from the visual, vestibular and somatosensorial systems in an integrated way to accurately regulate body positioning and center of mass movements. If one or more of these systems fail, or the sensory information is not correctly processed, the risk of a fall or instability increases. LBP can alter the sensory input to postural control ,hence leads towards lumbar instability due to weakness of core muscles in chronic low back pain it will leads to hypermobility of lumbar spine which will further adds to deterioration of internal homeostasis and motor control of lumbar spine. SEMG biofeedback can be used to help "down-train" elevated muscle activity or to "up-train" weak, inhibited, or paretic muscles.

This study will be Single blind Parallel group randomized controlled trial. The study settings will be Riphah College of Rehabilitation And Allied Health Sciences Lahore, Department of Physical Medicine and Rehabilitation Sciences, Fauji foundation Hospital Rawalpindi and Foundation University Institute of Rehabilitation Sciences. On Probability Purposive Sampling Technique will be used for sampling .A sample of 52 patients of mechanical low back pain will be obtained by using online sample calculator clincalc.com. Subjects will be randomized in to two groups i.e. Control group includes core stability exercises. Experimental group core stability with sEMG biofeedback using sealed envelope method with 1:1. In current study the assessor will be blinded from treatment allocation. The study participants satisfying the inclusion and exclusion criteria will be recruited in this trial after informed consent. Baseline assessment will be done on all participants by a Physical therapist Patients will be randomly allocated to control group (n=26), and interventional groups (n=26).Treatment will be given 3 times a week by researcher for 6 weeks with a total of 18 sessions for each patient .Re-assessment will then be done after 2nd week 4th week and at termination of treatment after 6th week

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders with mechanical low back pain
2. Patients with Lumbar Derangement Syndrome. (Mckenzie Classification)
3. Age: 18 to 60 years
4. Patients of both gender
5. NPRS ratings greater than 5
6. Constant or Intermittent pain worsening on repeated movements -

Exclusion Criteria:

1. Patients with non-mechanical low back pain
2. Patients with acute low back pain.
3. Post laminectomy/discectomy
4. Spondylolisthesis
5. Osteoporosis/Fractures
6. Cauda equine syndrome
7. Recent history of spinal trauma or surgery
8. Lumbar myelopathy
9. Patients with known metabolic diseases
10. Patients with any neurological deficit
11. Patients with any vestibular problems 12 Patients with visual impairment -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Postural Stability | 6 weeks
  it will be measured by using postural stability Balance System (R=0.94) (WJC Cachupe et al, 2001). This test is performed with open eyes as well as eyes closed and overall stability index will be calculated at the end of the test along with the percentage of time spent in each of the quadrants and zones (A to D).This test also provided information about the anterior /posterior index and Medial/Lateral index of participation

SECONDARY OUTCOMES:
Sensory integration of Balance | 6 weeks
  The Clinical Test of Sensory Interaction and Balance CTSIB is an accepted test protocol for sensory component of Balance assessment on a static surface. The CTSIB test protocol was selected for Fall Risk assessment as it is well documented in the literature as an effective test in identifying individuals with mild to severe balance problems Clinical test of Sensory Integration of Balance (CTSIB) using 4 different conditions using balance Balance System (R=0.94) (WJC Cachupe et al, 2001)
  * Eyes open firm surface: Baseline: Incorporates visual, vestibular and somatosensory inputs
  * Eyes closed firm surface: Eliminate visual input to evaluate vestibular and somatosensory inputs.
  * Eyes open on a dynamic surface used to evaluate somatosensory interaction with visually input
  * Eyes closed on dynamic surface: used to evaluate somatosensory interaction with vestibular input
Low Back Pain | 6 weeks
  Numerical pain rating scale is a patient self-report scale for measurement of pain intensity in the clinical and research settings. The NPRS has reliability from 0.67-0.96 patient rate his pain on the scale of 0-10: 0 - (no pain) and 10 - (worst pain).
Low back related functional disability | 6 weeks
  The Roland-Morris Disability Questionnaire is designed to assess self-rated physical disability caused by low back pain. The Roland-Morris Disability Questionnaire is most sensitive for patients with mild to moderate disability due to acute, sub-acute or chronic low back pain. (R= 0.42 - 0.91) Macedo et al. (2011)
Lumbar Range of Motion | 6 weeks
  Lumbar Physiological movements including forward bending, backward bending, and Right & Left side bending measured via Bubble Inclinometer. Inter-rater and intra-rater reliability for the inclinometer with Intra-class Correlation Coefficients of 0.90 and 0.85 for lumbar

CONTACTS AND LOCATIONS:
Overall Officials: Dr Rabiya Noor, Phd, Principal Investigator — Riphah University Lahore
Locations (2):
- Pakistan (2):
  - Foundation University Islamabad, Islamabad, Punjab Province
  - Riphah University Lahore, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No